CLINICAL TRIAL: NCT06811688
Title: The Effectiveness of Mobile Phone Reminders in the Improvement of Oral Hygiene in Patients With Fixed Orthodontic Appliances: A Randomized Controlled Trial
Brief Title: Effectiveness of Mobile Phone Reminder Applications in Improving Oral Hygiene Compliance of Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shahinaz N. Sembawa, Assistant Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAPO-02-K-012-2023-02-1459; +966125270000 (Other: Umm Al-Qura University)
Record Dates: First submitted 2025-01-23; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Oral Hygiene
Keywords: Active reminders; Mobile application; Oral hygiene; Orthodontic fixed appliance

STUDY DESIGN:
Intervention Model Description: The participants were asked to download two mobile applications: Brushout and Brush teeth reminder applications. These applications were adjusted to send notifications twice daily in the morning and night as reminders to practice oral hygiene.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal oral hygiene instructions group (No Intervention): Only verbal instructions on oral hygiene including brushing using soft bristles, brushing for 2 minutes, flossing once daily, the use of fluoridated oral rinse, orthodontic appliance care and avoiding hard and sticky food. These instructions were given at the baseline visit. Then, these subjects were re-examined after 4 weeks
- Smartphone reminder application group (Experimental): the subjects received the same oral hygiene instructions that were described to the control group with the addition of downloading two mobile applications: Brushout app and Brush teeth reminder app. These applications were adjusted to send notifications twice daily in the morning and night as reminders to practice oral hygiene. In addition, oral hygiene practice was tracked by a link that was sent electronically and checked by study researchers as a compliance protocol. Like the control group, subjects were re-examined after 4 weeks.
  Interventions: Other: Two mobile applications: Brushout and Brush teeth reminder applications

INTERVENTIONS:
Other: Two mobile applications: Brushout and Brush teeth reminder applications — These applications were adjusted to send notifications twice daily in the morning and night as reminders to practice oral hygiene.
  Other Names: reminder applications; mobile applications; smartphone application
  Arms: Smartphone reminder application group

SUMMARY:
The aim of this Randomized Controlled Trial (RCT) was to investigate the effectiveness of mobile application as an active reminder for improving oral hygiene compliance of patients undergoing orthodontic treatment using fixed orthodontic appliances.

DETAILED DESCRIPTION:
eligible participants will be randomly assigned to either control or intervention group. Group l (control): Only verbal instructions on oral hygiene including brushing using soft bristles, brushing for 2 minutes, flossing once daily, the use of fluoridated oral rinse, orthodontic appliance care and avoiding hard and sticky food.These instructions were given at the baseline visit. Then, these subjects were re-examined after 4 weeks. Group II (intervention): the subjects received the same oral hygiene instructions that were described to the control group with the addition of downloading two mobile applications: Brushout app and Brush teeth reminder app. These applications were adjusted to send notifications twice daily in the morning and night as reminders to practice oral hygiene. In addition, oral hygiene practice was tracked by a link that was sent electronically and checked by study researchers as a compliance protocol. Like the control group, subjects were re-examined after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

- 1- Subjects having orthodontic treatment using fixed appliances

2- The use of a smartphone to download Brushout app and Brush teeth reminder app

Exclusion Criteria:

* Subjects having orthodontic treatment using removable appliances

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Plaque Index | At baseline and 4 weeks
  As described by Silness-Löe plaque index, Six teeth (#16, #12, #24, #36, #32, #44) were used to evaluate the plaque present in each surface including facial, lingual, mesial and distal surface. The thickness of the plaque was measured as follows: 0: absence of microbial plaque, 1: thin film of microbial plaque along the free gingival margin, 2: moderate accumulation with plaque in sulcus, 3: large amount of plaque in sulcus or pocket along the free gingival margin.
Gingival index | At baseline and 4 weeks
  Gingival index was used to evaluate the gingival condition in each surface including facial, lingual, mesial and distal. The following scores were used: 0: normal gingiva 1: mild inflammation- slight change in color, slight edema and no bleeding on probing, 2: moderate inflammation- redness, edema and glazing and bleeding on probing 3: severe inflammation- marked redness and edema and tendency to spontaneous bleeding, ulceration.

CONTACTS AND LOCATIONS:
Overall Officials: Shahinaz N Sembawa, PhD, Principal Investigator — Umm AlQura University
Locations (1):
- Umm Al-Qura University, Dental Teaching Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jepsen K, Sculean A, Jepsen S. Complications and treatment errors involving periodontal tissues related to orthodontic therapy. Periodontol 2000. 2023 Jun;92(1):135-158. doi: 10.1111/prd.12484. Epub 2023 Mar 15. PMID 36920050
- [Background] Santonocito S, Polizzi A. Oral Microbiota Changes during Orthodontic Treatment. Front Biosci (Elite Ed). 2022 Jul 27;14(3):19. doi: 10.31083/j.fbe1403019. PMID 36137992
- [Background] Patil S, Hedad IA, Jafer AA, Abutaleb GK, Arishi TM, Arishi SA, Arishi HA, Jafer M, Gujar AN, Khan S, Raj AT. Effectiveness of mobile phone applications in improving oral hygiene care and outcomes in orthodontic patients. J Oral Biol Craniofac Res. 2021 Jan-Mar;11(1):26-32. doi: 10.1016/j.jobcr.2020.11.004. Epub 2020 Nov 17. PMID 33344158
- [Background] Pascadopoli M, Zampetti P, Nardi MG, Pellegrini M, Scribante A. Smartphone Applications in Dentistry: A Scoping Review. Dent J (Basel). 2023 Oct 20;11(10):243. doi: 10.3390/dj11100243. PMID 37886928